CLINICAL TRIAL: NCT00802594
Title: Phase II A Trial of DB289 for the Treatment of Stage I African Trypanosomiasis
Brief Title: A Trial of DB289 for the Treatment of Stage I African Trypanosomiasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Immtech Pharmaceuticals, Inc (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Christian Burri, MSc, PhD., Swiss Tropical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 289-C-003
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-12

CONDITIONS: Trypanosomiasis, African
Keywords: first stage; T.b. gambiense; sleeping sickness; Patients with first stage T.b. gambiense sleeping sickness
MeSH Terms: conditions — Trypanosomiasis, African

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DB289 (Experimental)
  Interventions: Drug: DB289

INTERVENTIONS:
Drug: DB289 — A single 100 mg DB289 capsule will be taken by mouth twice a day, morning and evening. Drug is to be taken with a glass of water within 15 minutes of the completion of meal.
  Other Names: pafuramidine maleate

SUMMARY:
Human African Trypanosomiasis or sleeping sickness has made a spectacular return during the last decade, and in many places the demand largely surpasses the capacities of the treatment centers. Treatment of the disease remains unsatisfactory. All currently used drugs must be administered parenterally, treatment is lengthy, and adverse drug reactions frequent. There are currently no drugs which might be used as a tool to support disease control that is easily administered and has low toxicity.

This study aims to assess the efficacy of DB289, a new, oral drug for treatment of first stage sleeping sickness. The project will be executed in the framework of an international consortium consisting of more than a dozen partners from academia, industry, and the Ministries of Health of Angola and the Democratic Republic of Congo.

DETAILED DESCRIPTION:
This is a single-center, open label, non-controlled Phase IIa trial. Patients with first stage T.b. gambiense sleeping sickness will receive 100 mg of DB289 orally twice a day for 5 days. Subjects meeting entry criteria will be enrolled at a single site.

A total of 30 patients will be enrolled in this trial. Enrollment is planned to begin third quarter 2001 and be completed in 2-3 months.

The study will be conducted at the Trypanosomiasis Reference Center, Viana (ICCT), Angola, and at the Trypanosomiasis Treatment Center in Maluku, Congo.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has early stage T. b. gambiense infection i.e. parasitologically confirmed infection in the blood or lymph and less than or equal to 5 WBC mm-3 detected in the CSF by microscopic examination
2. Patient is 16 years old or more
3. Patient has a minimal weight of 45 kilograms
4. If patient is female of child bearing potential (a women will be considered of non-child bearing potential only if she has been post menopausal for over 2 years or has had a hysterectomy), she is not lactating, she had a negative urine pregnancy test result within 24 hours prior to DB289 treatment and she agrees to use a medically proven method of contraception (abstinence from sexual intercourse acceptable) from the day of consent on until 7 Days after DB289 treatment completion (Study Day 12).
5. Patient has signed the Informed Consent. If the patient is minor, a legal guardian has signed the Informed Consent

Exclusion Criteria:

1. The patient has late stage T.b. gambiense infection i.e. presence of parasite in the CSF upon microscopic examination, or a positive (titer greater than 1/4) latex / IgM test, or a positive latex / T.b.g.
2. Active clinically relevant medical conditions that in the Investigator opinion may jeopardize subject safety or interfere with participation in the study, including but not limited to: significant liver diseases, chronic pulmonary diseases, significant cardiovascular diseases or significant ECG anomaly such as elongated QTc (corrected) interval above 430 msec for men or above 450 msec for women, diabetes, thyroid diseases, gout, infection including known HIV infection, CNS trauma or seizure disorders.
3. Clinically significant abnormal laboratory value at screening including:

   * Prothrombin Time > 1.25 times upper limit of normal (ULN)
   * Liver enzyme AST and ALT > 2 times ULN
   * Total bilirubin > 1.5 times ULN
   * Serum Creatinine > 1.5 times ULN
4. Traumatic lumbar puncture (i.e. red blood cells visible in CSF)
5. Coma Score of less than 9 on the Glasgow Coma Scale (Appendix 8)
6. Withdrawal of consent at any time during the study
7. Any condition which compromises ability to communicate with the investigator as required for the completion of this study.
8. The subject has been previously treated for African Trypanosomiasis.
9. The subject has been previously enrolled in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2001-08; Primary Completion 2002-08 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the parasitological cure 24 hours after completion of treatment. | Day 7
The primary outcome measure for safety analysis will be the rate of occurrence of Grade 3 or higher adverse events during the observation period. | Day 12

SECONDARY OUTCOMES:
A secondary endpoint is the parasitological cure 3, 6, 12, 24 months after completion of treatment. | 3, 6, 12, 24 months
The secondary outcome measure will be the incidence rate of adverse events (all Grades combined) during the observation period (as compared to literature values for pentamidine). | Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Christian Burri, MSc, PhD, Study Director — Swiss Tropical & Public Health Institute
Locations (2):
- Laboratory of Reference and Investigation, Viana, ICCT, Bairro Ingombota, Luanda Province, Angola
- Programme National de Lutte contre la Trypanosomiase, Kinshasa, Gombe, Republic of the Congo

REFERENCES:
- [Derived] Burri C, Yeramian PD, Allen JL, Merolle A, Serge KK, Mpanya A, Lutumba P, Mesu VK, Bilenge CM, Lubaki JP, Mpoto AM, Thompson M, Munungu BF, Manuel F, Josenando T, Bernhard SC, Olson CA, Blum J, Tidwell RR, Pohlig G. Efficacy, Safety, and Dose of Pafuramidine, a New Oral Drug for Treatment of First Stage Sleeping Sickness, in a Phase 2a Clinical Study and Phase 2b Randomized Clinical Studies. PLoS Negl Trop Dis. 2016 Feb 16;10(2):e0004362. doi: 10.1371/journal.pntd.0004362. eCollection 2016 Feb. PMID 26881924